CLINICAL TRIAL: NCT04039828
Title: Zinc Sulfate Acceptability Study in Children With Acute Diarrhea: A Prospective, Open-label, Interventional Study
Brief Title: Zinc Sulfate Acceptability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-19033
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2019-07

CONDITIONS: Acute Diarrhea
Keywords: Diarrhea; 3 to 59 months children; Zinc tablet; acceptability; adherence; palatability
MeSH Terms: conditions — Diarrhea | interventions — Zinc Sulfate; Tablets; Zinc

STUDY DESIGN:
Intervention Model Description: Stratum 1: From 3 months to <18 months= 175 Stratum 2: From 18 months to 59 months= 175
  in total, 350 participants will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stratum (Experimental): Stratum 1: From 3 months to <18 months= 175 Stratum 2: From 18 months to 59 months= 175
  In total, 350 participants will be enrolled
  Interventions: Drug: Zinc Sulfate Dispersible Tablet 20 mg (Elemental Zinc 20 mg as Zinc Sulfate Monohydrate / Tablet)

INTERVENTIONS:
Drug: Zinc Sulfate Dispersible Tablet 20 mg (Elemental Zinc 20 mg as Zinc Sulfate Monohydrate / Tablet) — Half of the tablet (10 mg) for 3 to 6 months old children and one tablet (20 mg) daily for > 6 to 59 months old children. The tablet will be dissolved in a teaspoon of safe water or breast milk and administered once daily for 10 days.
  Other Names: Zinc, Zinc dispersible tablet

SUMMARY:
Introduction:

Zinc (Zn) is an essential mineral widely distributed within the human body with metalloproteins, Zinc-binding proteins, etc. It is necessary for signal transduction and also cell growth and proliferation via respective metallo- and zinc-dependent enzymes. Zinc supplementation can significantly reduce diarrheal severity and duration as well as prevents future incidences and reduces use of other medications in diarrhoea. For this reason WHO, UNICEF, USAID and experts worldwide jointly recommended zinc supplementation (10 mg for infants less than 6 months old and 20 mg in 6 - 59 months old) combined with reduced osmolarity ORS for clinical management of acute diarrhoea. But due to strong metallic taste zinc products are less palatable to children even after using masking flavours as recommended by WHO. Several companies have formulated the product since WHO recommendations came but still transient side effects like vomiting and regurgitation remain evident. Despite careful counselling to the caregivers expected adherence rate to 10 days regimen of zinc supplement is yet to be reached.

With the aim to increase zinc supplement coverage during acute diarrheal illness, it is necessary to conduct a study to introduce new formulation Zinc tablet which is more palatable, more dispersible and more acceptable.

Intervention:

Zinc sulfate [Zinc Dispersible Tablet, 20 mg; (Elemental Zinc 20 mg as Zinc Sulfate Monohydrate / Tablet)]

Methods: Prospective, open label, interventional study

Hypothesis:

Improved formulation of Zinc Sulfate will have good acceptability.

Study population:

Stratum 1: 3 months - <18 months = 175 children Stratum 2: 18 months - 59 months = 175 children

Objectives:

1. Primary Objective:

   Acceptability of the zinc product in the management of childhood diarrhea will be assessed by observing:

   i) Incidence of vomiting or regurgitation among enrolled children receiving the improvised zinc formulation.

   ii) The adherence: The number of days (out of the total 10 days) the child took the protocol-prescribed dose of the medicine. The treatment will be considered to have good acceptability if at least 80% of the prescribed treatment is taken by at least 70% of the children over the duration of 10 days, as per WHO guidelines.
2. Secondary objective :

To assess palatability Secondary end point evaluation (Palatability): The statistical analysis will comprise the calculation of the percentage of patients out of 350 who found the investigational product to have "very well-tolerated, well-tolerated or tolerated" scores (i.e. any of the upper 3 possible scores). A 95% confidence interval, using the normal approximation of the binomial distribution, will be calculated for the percentage.

DETAILED DESCRIPTION:
Background:

Zinc is a metalloprotein. The two important function of zinc are- first, unlike other metals zinc is virtually non-toxic (1). The homeostatic mechanisms that regulate its entrance, allocation, and excretion from cells and tissues are so well-organized that no disorders are known to be associated with its excessive accumulation, in contrast to iron, copper, mercury, and other metals. Second, its physical and chemical properties, including its generally stable relationship with macromolecules and its co-ordination flexibility, make it extremely adaptable in meeting the needs of proteins and enzymes that take diverse biological functions (2-4). Zinc is one of the most common metal ion distributed widely in cytoplasm as well as building blocks for keratin like structures and intracellular organelles like chromosomes(5). Importance of zinc as an essential trace element is well established for its role on growth and development, protection against free radical damage, endocrine, reproductive and cognitive functions(6). Globally, zinc deficiency is associated with 16% of lower respiratory tract infections and 10% of diarrheal diseases respectively with higher attributable fractions in sub-regions(7). Severe zinc deficiency is a rare entity whereas mild to moderate zinc deficiency is quite evident mostly in children living in poverty and associated with approximately 453,000 deaths each year(8, 9). Simultaneously, diarrhoea as the second most prevalent cause of under five deaths and is responsible for 800,000 deaths each year (10). A meta-analysis of 12 studies observed the impact of zinc supplements on the management of acute diarrhea, 11 studies showed a reduction in the duration of the diarrheal episode. In eight of these reported that the reduction of diarrheal episode was statistically significant. Five of these studies also found that zinc supplements reduced stool output and frequency. The data revealed that zinc supplementation had a significant effect on the clinical course of acute diarrhea, reducing its duration as well as severity (11). Another meta-analysis of 18 trials with 6165 enrolled participants observed that in acute diarrhea, zinc reduced duration of diarrhea (MD -- 12.27 hours, 95% CI -23.02 to -1.52 hours; 2741 children, nine trials), and a reduced amount of diarrhea by day three (RR 0.69, 95% CI 0.59 to 0.81; 1073 children, two trials), day five (RR 0.55, 95% CI 0.32 to 0.95; 346 children, two trials), and day seven (RR 0.71, 95% CI 0.52 to 0.98; 4087 children, seven trials). Zinc also reduced the period of persistent diarrhea (MD -15.84 hours, 95% CI -25.43 to - 6.24 hours; 529 children, five trials). In few trials there was report on the severity, but the results were not consistent (12).

Zinc supplementation can significantly reduce diarrheal severity and duration as well as prevents future incidences and reduces use of other medications in diarrhea (13-16). Several studies evaluated the effect of zinc supplementation on diarrhea and found a preventive and long-lasting impact. These showed that 10 mg to 20 mg of zinc per day, for 10 - 14 days, reduced the number of diarrheal episodes in 2 - 3 months after the supplementation (12). For this reason WHO, UNICEF, USAID and experts worldwide jointly recommended zinc supplementation (10 mg for infants less than 6 months old and 20 mg in 6 - 59 months old) combined with reduced osmolarity ORS for clinical management of acute diarrhoea (17).

The physiological effect of zinc on intestinal ion transport has not yet been established thoroughly. In in-vitro studies with rat ileum recently established that zinc inhibits cAMP-induced, chloride-dependent fluid secretion by inhibiting basolateral potassium (K) channels. This study has also observed the specificity of Zn to cAMP-activated K channels, because zinc did not block the calcium (Ca)-mediated pottasium channels. As this study was not done in Zn-deficient animals, it provides support that Zn is probably effective in the absence of Zn deficiency (18, 19). Zinc also improves the absorption of water and electrolytes, improves regeneration of the intestinal epithelium, increases the levels of brush border enzymes, and enhances the immune response, allowing for a better clearance of the pathogens. Another report has recently shown evidence that zinc inhibits toxin-induced cholera, but not Escherichia coli heat-stable, enterotoxin-induced, ion secretion in cultured Caco-2 cells (20). In this way, Zinc plays an important role in modulating the host resistance to infectious agents and decreases the risk, severity, and duration of diarrheal diseases. It also plays an important role in metallo-enzymes, polyribosomes, and the cell membrane and cellular function, giving belief that it plays a central role in cellular growth and in the function of the immune system (21).

The primary site of absorption of exogenous zinc in the human is in the proximal small bowel, either the distal duodenum or proximal jejunum ((22). Factors known to control absorption include the amount of zinc present in the intestinal lumen, the presence of dietary promoters (e.g., human milk, animal proteins) or inhibitors (e.g., phytate, other minerals), zinc "status" especially in relation to chronic zinc intake, and physiologic states (23).

After absorption zinc is bound to protein metallothionein in the intestines. Zinc is widely distributed throughout the body. It is primarily stored in RBCs, WBCs, muscles, bones, Skin, Kidneys, Liver, Pancreas, retina, and prostate. The extent of Zinc binding is 60 - 70% to plasma albumin, 30 - 40% to alpha 2 macroglobulins or transferring, and 1% to amino acids like histidine and cysteine. Peak plasma concentration of Zinc occurs in approximately two hours. The processes of secretion and reabsorption or excretion of intestinal endogenous zinc have not been well characterized in humans. There are several potential sources of the endogenous zinc: pancreatic and biliary secretions, gastroduodenal secretions, transepithelial flux from the enterocytes or other intestinal cell types and sloughing of mucosal cells.(23) Zinc sulfate, acetate, and gluconate are all acceptable zinc salt formulations, of which zinc sulfate is low-cost, efficacious, safe, and therefore, optimal for the national program. Zinc sulfate tablets may be dispersed in breast milk, in oral rehydration solutions, or in water on a small spoon. Zinc sulfate dispersible tablet is also available in the market, containing 20 mg of elemental zinc. Pediatric zinc sulfate tablets are also available(24) It has been anticipated that the successful scaling up of zinc supplementation for childhood diarrhea could potentially save 400,000 under-five deaths per year (25). The Scaling Up of Zinc for Young Children (SUZY) Project was established in 2003 with the aim of setting Bangladesh on the path to covering all under-five children with zinc supplementation in any diarrheal illness episode. In December, 2006 a national mass media campaign to promote a dispersible tablet zinc formulation, "Baby Zinc," for management of childhood diarrhea was launched. All media messages linked zinc treatment to the continued use of oral rehydration salts (ORS)(26). However, by 2012, zinc coverage was below 5% globally though in some countries such as Bangladesh, coverage was as high as 41% (27). According to WHO, Bangladesh was the only country to achieve high treatment rates nationally: as of 2014 nearly 80% of children with diarrhea received ORS, and 34% received both ORS and zinc (28). This was achieved through decades of investment by the government, icddr,b, the international development organizations, BRAC, and other key stakeholders (29, 30). This endeavor included the large-scale Scaling Up Zinc for Young Children (SUZY) Project which was initiated in 2003 and included partnerships with the government, non-governmental organizations (NGOs), the private sector to improve provider dispensing, caregiver demand and availability of optimal, affordable products (26, 31).

But combined data collected from five RCTs (n = 3156) observed that zinc significantly increased the chance of vomiting compared to the control agent (RR1.2, 95% CI 1.05-1.4)(32). Due to strong metallic taste zinc products are less palatable to children even after using masking flavours as recommended by WHO. Several companies have formulated the product since WHO recommendations came but still transient side effects like vomiting and regurgitation remain evident (33-36). Despite careful counselling to the caregivers expected adherence rate to 10 days regimen of zinc supplement is yet to be reached (33, 35, 37, 38).

A clinical trial with new formulation Zinc Sulfate for use in acute diarrheal illness will be conducted to achieve good adherence rate. New improvised Zinc preparation will be palatable, more dispersible and thereby acceptable to young children with diarrhea.

Study design: Prospective, open label, interventional study

Study Site: The study will be conducted at the Dhaka Hospital of the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b).

Study population:

Stratum- I : 3 months - <18 months Stratum- II : 18 months - 59 months

Sample size:

Sample size is estimated considering the primary outcome variables:

For one component of the primary objective we have considered the study-report done by Khan et al (34), where they found incidence of vomiting or regurgitation in 22% of enrolled children. We assume that the incidence of vomiting or regurgitation on receiving the improvised zinc formula would not be greater than 10 % cases in this study, thus a total 300 children will be needed that would accommodate up to 19% attrition. Sample size is calculated using the formula [ 2(Zα + Zβ)2 * p * q] / d2

Where:

P = (p1+p2)/2 p1 = 22% incidence of vomiting or regurgitation according to study report done by Khan et al p2 = 10% incidence of vomiting or regurgitation with the improvised zinc formula that we are assuming Zα = 5% significance level Zβ = (1 -β) = 80% power p = [p1 (22%) + p2 (10% )]/2 = 16%; q = 100% -16% = 84%; Zα = 1.96 and Zβ = 1.64 Sample size is further estimated for the other component of the primary objective, i.e. adherence. A total of 350 children will be enrolled (175 patients from 3 months to below 18 months age group, and 175 children from 18 months to 59 months age group). To identify a ± 7.5% minimal difference in acceptability between children aged over and below 18 months with an anticipated 70% acceptability (p), setting the level of confidence at 95% (z = 1.96) using the formula: pqz2/ d2 the estimated sample size is 175 children per group allowing 18% dropout.

Intervention:

Investigational product: Zinc Sulfate [Zinc Dispersible Tablet, 20 mg; (Elemental Zinc 20 mg as Zinc Sulfate Monohydrate / Tablet)]

Dosage:

Half the tablet (10 mg) for 3 to 6 months old children and 20 mg daily for > 6 to 59 months old children. The tablet will be dissolved in a teaspoon of safe water or breast milk and administered once daily for 10 days.

Packaging and labeling: Investigational product will be dispensed in a blister pack containing 10 tablets.

The caregivers will bring the blister packs (even if all tablets are used) on day 11 (after enrollment) for a follow up visit to the outpatient department (OPD) of the Dhaka Hospital of icddr,b, and they will be evaluated about the adherence with the supplied drug intake during the follow up visit. Study investigator will update accountability records of the investigational product according to ICH E6, GCP guideline. If caregiver failed to have the follow up visit at hospital, the study staff will visit children's house after 12 days of enrollment. Investigational product will not be provided to any third party.

References:

1. Seiler HG, Sigel H, Sigel A. Handbook on toxicity of inorganic compounds. 1988.
2. Vallee BL, Auld DS. Zinc coordination, function, and structure of zinc enzymes and other proteins. Biochemistry. 1990;29(24):5647-59.
3. Vallee BL, Auld DS. Short and long spacer sequences and other structural features of zinc binding sites in zinc enzymes. FEBS letters. 1989;257(1):138-40.
4. Vallee BL, Auld DS. Active-site zinc ligands and activated H2O of zinc enzymes. Proceedings of the National Academy of Sciences. 1990;87(1):220-4.
5. Mills CF. Zinc in human biology: Springer Science & Business Media; 2013.
6. Organization WH. Trace elements in human nutrition and health. 1996.
7. McCall KA, Huang C-c, Fierke CA. Function and mechanism of zinc metalloenzymes. The Journal of nutrition. 2000;130(5):1437S-46S.
8. Prasad AS. Zinc deficiency in human subjects. Progress in clinical and biological research. 1983;129:1-33.
9. Walker CF, Ezzati M, Black R. Global and regional child mortality and burden of disease attributable to zinc deficiency. European journal of clinical nutrition. 2009;63(5):591.
10. UNICEF. Diarrhoea remains a leading killer of young children, despite the availability of a simple treatment solution. UNICEF Data: Monitoring the Situation of Children and Women. 2016. 2018.
11. Organization WH. Clinical management of acute diarrhoea: WHO. Geneva: World Health Organization, 2004.
12. LAZZERINI M, GRAY D. Oral zinc for treating diarrhoea in children. Commentary. International journal of epidemiology. 2008;37(5):938-40.
13. Bhutta Z, Black RE, Brown K, Gardner JM, Gore S, Hidayat A, et al. Prevention of diarrhea and pneumonia by zinc supplementation in children in developing countries: pooled analysis of randomized controlled trials. The Journal of pediatrics. 1999;135(6):689-97.
14. Baqui AH, Black RE, El Arifeen S, Yunus M, Chakraborty J, Ahmed S, et al. Effect of zinc supplementation started during diarrhoea on morbidity and mortality in Bangladeshi children: community randomised trial. Bmj. 2002;325(7372):1059.
15. Strand TA, Chandyo RK, Bahl R, Sharma PR, Adhikari RK, Bhandari N, et al. Effectiveness and efficacy of zinc for the treatment of acute diarrhea in young children. PEDIATRICS-SPRINGFIELD-. 2002;109(5):898-903.
16. Group ICZEfD. Zinc supplementation in acute diarrhea is acceptable, does not interfere with oral rehydration, and reduces the use of other medications: a randomized trial in five countries. Journal of pediatric gastroenterology and nutrition. 2006;42(3):300-5.
17. UNICEF Wa. WHO/UNICEF Joint Statement: Clinical management of acute diarrhoea, WHO, Geneva, 2004 2004. Available from: http://www.unicef.org/publications/files/ENAcute_Diarrhoea_reprint.pdf.
18. Hoque KM, Rajendran VM, Binder HJ. Zinc inhibits cAMP-stimulated Cl secretion via basolateral K-channel blockade in rat ileum. American Journal of Physiology-Gastrointestinal and Liver Physiology. 2005;288(5):G956-G63.
19. Hoque KM, Binder HJ. Zinc in the treatment of acute diarrhea: current status and assessment. Gastroenterology. 2006;130(7):2201-5.
20. Canani RB, Cirillo P, Buccigrossi V, Ruotolo S, Passariello A, De Luca P, et al. Zinc inhibits cholera toxin-induced, but not Escherichia coli heat-stable enterotoxin-induced, ion secretion in human enterocytes. The Journal of infectious diseases. 2005;191(7):1072-7.
21. Organization WH, UNICEF. Implementing the new recommendations on the clinical management of diarrhoea: guidelines for policy makers and programme managers. 2006.
22. Krebs N, Westcott J, Huffer J, Miller L, editors. Absorption of exogenous zinc (Zn) and secretion of endogenous Zn in the human small intestine. FASEB JOURNAL; 1998: FEDERATION AMER SOC EXP BIOL 9650 ROCKVILLE PIKE, BETHESDA, MD 20814-3998 USA.
23. Krebs NF. Overview of zinc absorption and excretion in the human gastrointestinal tract. The Journal of nutrition. 2000;130(5):1374S-7S.
24. Stuart MC, Kouimtzi M, Hill SR. WHO model formulary 2008: World Health Organization; 2009.
25. Jones G, Steketee RW, Black RE, Bhutta ZA, Morris SS, Group BCSS. How many child deaths can we prevent this year? The lancet. 2003;362(9377):65-71.
26. Larson CP, Saha UR, Nazrul H. Impact monitoring of the national scale up of zinc treatment for childhood diarrhea in Bangladesh: repeat ecologic surveys. PLoS medicine. 2009;6(11):e1000175.
27. Unger CC, Salam SS, Sarker MSA, Black R, Cravioto A, El Arifeen S. Treating diarrhoeal disease in children under five: the global picture. Archives of disease in childhood. 2014;99(3):273-8.
28. Calverton M. National Institute of Population Research and Training (NIPORT). Mitra and Associate and ORC Macro. 2005.
29. Chowdhury AMR, Karim F, Sarkar S, Cash RA, Bhuiya A. The status of ORT in Bangladesh: how widely is it used? Health Policy and Planning. 1997;12(1):58-66.
30. Mosites E, Hackleman R, Weum K, Pintye J, Manhart J, Hawes SE. Bangladesh ORS case study. Seattle, WA: Bill & Melinda Gates Foundation and University of Washington Global Health START Program. 2012.
31. Larson CP, Koehlmoos TP, Sack DA, Team SUoZfYCP. Scaling up zinc treatment of childhood diarrhoea in Bangladesh: theoretical and practical considerations guiding the SUZY Project. Health policy and planning. 2011;27(2):102-14.
32. Patro B, Golicki D, Szajewska H. Meta-analysis: zinc supplementation for acute gastroenteritis in children. Alimentary pharmacology & therapeutics. 2008;28(6):713-23.
33. Ahmed S, Nasrin D, Ferdous F, Farzana FD, Kaur G, Chisti MJ, et al. Acceptability and compliance to a 10-Day regimen of zinc treatment in diarrhea in rural Bangladesh. Food and Nutrition Sciences. 2013;4(04):357.
34. Khan AM, Larson CP, Faruque AS, Saha UR, Hoque AB, Alam NU, et al. Introduction of routine zinc therapy for children with diarrhoea: evaluation of safety. J Health Popul Nutr. 2007;25(2):127-33.
35. Nasrin D, Larson CP, Sultana S, Khan TU. Acceptability of and adherence to dispersible zinc tablet in the treatment of acute childhood diarrhoea. J Health Popul Nutr. 2005;23(3):215-21.
36. Larson CP, Hoque AB, Larson CP, Khan AM, Saha UR. Initiation of zinc treatment for acute childhood diarrhoea and risk for vomiting or regurgitation: a randomized, double-blind, placebo-controlled trial. J Health Popul Nutr. 2005;23(4):311-9.
37. Lamberti LM, Walker CLF, Taneja S, Mazumder S, Black RE. Adherence to zinc supplementation guidelines for the treatment of diarrhea among children under-five in Uttar Pradesh, India. Journal of global health. 2015;5(2).
38. Valekar SS, Fernandez K, Chawla P, Pandve H. Compliance of zinc supplementation by care givers of children suffering from diarrhea. Indian Journal of Community Health. 2014;26(Supp 2):137-41.
39. Alam NH, Ashraf H. Treatment of infectious diarrhea in children. Pediatric Drugs. 2003;5(3):151-65.
40. Patel A, Mamtani M, Dibley MJ, Badhoniya N, Kulkarni H. Therapeutic value of zinc supplementation in acute and persistent diarrhea: a systematic review. PLoS One. 2010;5(4):e10386.
41. Lukacik M, Thomas RL, Aranda JV. A meta-analysis of the effects of oral zinc in the treatment of acute and persistent diarrhea. Pediatrics. 2008;121(2):326-36.
42. Therapeutic effects of oral zinc in acute and persistent diarrhea in children in developing countries: pooled analysis of randomized controlled trials-. The American journal of clinical nutrition. 2000;72(6):1516-22.
43. Haider BA, Bhutta ZA. The effect of therapeutic zinc supplementation among young children with selected infections: a review of the evidence. Food and nutrition bulletin. 2009;30(1_suppl1):S41-S59.

ELIGIBILITY:
Inclusion Criteria:

* Children of age 3 - 59 months with an acute diarrhea episode who will be prescribed oral re-hydration salts (ORS) per WHO guidelines
* Residence: within 10 km of the Dhaka Hospital of icddr,b
* Signed informed consent by the guardians/caregivers

Exclusion Criteria:

* Some or severe dehydration
* Already in the middle of a course of zinc sulfate due a recent previous episode
* Severe acute malnutrition (weight for height < - 3 z score or bi-pedal edema)
* Congenital anomalies
* Fever or invasive diarrhea or any other medical illness (other than acute diarrhea)
* Having any known medical condition that may interfere with the subject's ability to sense or discriminate between different tastes

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 325 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of the Zinc Dispersible Tablet | Adherence will be measured on 11th day after enrollment (Following 10 days regimen of investigational Zinc Dispersible Tablet).
  The treatment will be considered to have good acceptability if 80% of the prescribed treatment is taken by at least 70% of the children.

SECONDARY OUTCOMES:
Taste palatability of Zinc Dispersible Tablet | Individual daily recorded responses (For 10 days during the drug administration) will be used to arrive at the overall response value on the 5-point pictorial Hedonic scale.
  A subjective evaluation measured on the basis of a caregiver's report of his/her child's behavior (through a 5-point pictorial Hedonic scale) during the 10 days when the medicine is administered. A 'Diary Card' will be provided to the caregiver for keeping the daily records of the events.

CONTACTS AND LOCATIONS:
Overall Officials: Azharul Islam Khan, PhD, MBBS, Principal Investigator — Chief Physician and Head, Hospitals, icddr,b
Locations (2):
- Bangladesh (2):
  - Dhaka Hospital, Dhaka
  - International centre for Diarrhoeal Disease Research, Bangladesh, Dhaka

REFERENCES:
- [Derived] Alam J, Nuzhat S, Billal SM, Ahmed T, Khan AI, Hossain MI. Nutritional Profiles and Zinc Supplementation among Children with Diarrhea in Bangladesh. Am J Trop Med Hyg. 2023 Feb 27;108(4):837-843. doi: 10.4269/ajtmh.22-0532. Print 2023 Apr 5. PMID 36848897